CLINICAL TRIAL: NCT07291973
Title: A Clinical Investigation in lUng canceR of the Endowave FlexAblate™ Microwave tRansbronchial Ablation System.
Brief Title: Clinical Investigation Evaluating the Performance, Safety and Clinical Benefit of the Endowave FlexAblate™ Microwave Ablation System in Patients Undergoing Lung Ablation Procedures.
Acronym: AURORA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endowave Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EDW-CID-001
Record Dates: First submitted 2025-11-25; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Microwave Ablation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, non-randomised clinical investigation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transbronchoscopic Microwave Ablation (Experimental): The FlexAblate™ Microwave Ablation System is deployed and used to conduct bronchoscopic ablations in the lung.
  Interventions: Device: Microwave Ablation

INTERVENTIONS:
Device: Microwave Ablation — FlexAblate Microwave Transbronchial Ablation System

SUMMARY:
The goal of this clinical trial is to learn if the FlexAblate™ Ablation System works to treat a lung cancer nodules and it will also learn about the safety of the ablation system.

Participants in this clinical trial will be patients aged over 18 years who have been previously diagnosed with cancer in the lung (primary or secondary malignant tumours) and deemed unsuitable for surgery or are declining surgery or, patients suitable for microwave ablation procedure based on clinical assessment.

Those who meet all of the eligibility criteria at a screening assessment (a review of eligibility to participate in the study includes review of information on the cancerous nodule, recording your medical history, current medications, a blood test, and quality of life assessments) will undergo the ablation treatment with FlexAblate™ Microwave Ablation System. Follow-up assessments will be at week 1 and months 1, 3, 6 and 12 will includes CT Scans (CT or "CAT" scan is a computed tomography scan), blood tests, assessment of overall health and quality of life assessments.

DETAILED DESCRIPTION:
This is a prospective, single-arm, non-randomised clinical investigation. Up to 43 subjects will be enrolled from up to 5 sites. The clinical investigation is designed to evaluate the performance and safety of the Endowave FlexAblate™ Microwave Ablation System device in subjects undergoing lung ablation procedures. Microwave Ablation System device in subjects undergoing lung ablation procedures.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years of age who has provided signed informed consent.
* Subject is able and willing to comply with the planned clinical investigation follow-up schedule
* Pathological confirmed malignant nodule in the lung either primary or metastatic disease.
* Target nodule is ≤ 20mm in maximum diameter.
* There is ≥ 5mm of nodule-free lung parenchyma between target nodule and pleura or fissure.
* Subject is a candidate for an elective lung ablation procedure as determined by institutional multi-disciplinary board or equivalent.
* Subject or the lesion is not suitable for surgery or patient refuses surgery.

Exclusion Criteria:

* Target nodule is abutting main or lobar stem bronchus, main pulmonary vasculature (vessel 5mm), heart, oesophagus and/or trachea.
* Subjects who are extremely breathless or on home oxygen therapy.
* Female subjects who are pregnant or nursing.
* Subjects with uncorrectable coagulopathy or thrombocytopenia at time of screening.
* Subjects with prior pneumonectomy.
* Subjects who have had any radiation (i.e., SBRT or EBRT) to the intended ablation zone or lung ablation, surgical resection therapy, radiotherapy, or any other treating procedure within 30 days prior to the planned ablation procedure or those who plan to receive a lung ablation, surgical resection, or radiation therapy on the ablated lung side before completing the primary endpoint assessment (30 days post-ablation).
* Subjects who have implantable electronic devices, including pacemakers or other electronic implants.
* Known pulmonary hypertension (Pulmonary artery systolic pressure, PASP >50mmHg).
* Active active pulmonary infection at time of screening or the procedure.
* Subjects medically unable to stop anticoagulant or anti-platelet therapy for relevant time period prior to and following the ablation procedure.
* Participation in an investigational drug or device clinical investigation within 30 days of enrolment that would interfere with this clinical investigation.
* The investigator determines that participation in this clinical investigation may jeopardise the safety or welfare of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical Efficacy | 1 month
  Technical Efficacy defined as ablation of the target tumour with the ablation zone completely overlapping or encompassing the entire target tumour assessed using conventional CT imaging.

SECONDARY OUTCOMES:
Procedure Technical Success | Day of procedure
  Procedure technical success defined by the investigator as successful deployment, activation and removal of the ablation catheter according to the investigation plan.
Ablation Technical Success | At Discharge - Day 1
  Ablation technical success defined as the nodule treated according to the investigation plan and covered completely by the ablation zone with an adequate margin assessed using CT imaging.
Safety Assessment - number of device or procedure related Serious Adverse Events | Through to 1 month follow-up
  Number of Serious Adverse events (SAE) related to the device or procedure associated with the use of the FlexAblate System.
Safety Assessment - number of device or procedure related Adverse Events (AE) | Through to 3 months
  Number of Adverse Events (AE) related to the device or procedure.
Quality of Life Assessment - European Organization for Research and Treatment of Cancer Quality of life questionnaire - Cancer (EORTC QLQ-C30) | 12 months
  Patients will rate their responses from 1 to 4 on a Likert Scale (1 being "not at all" and 4 being "very much").
Quality of Life Assessment - EQ-5D-5L health-related quality of life questionnaire | 12 months
  Patients complete the 5 level descriptive system relating to 5 dimensions of health and the EQ visual analogue scale from 0 to 100 (where 0 means the worst health you can imagine and 100 means the best health you can imagine).
Quality of Life Assessment - Bronchoscopic Ablation Patient Pain and Satisfaction Survey | 1 month
  Survey completed by the patient to assess their pain and satisfaction with the ablation procedure.

OTHER OUTCOMES:
Ablation zone size assessment | Discharge - Day 1
  Evaluation of the ablation zone size defined as the radiologic region or zone of induced treatment effect by CT imaging.
Assessment of Local Control | 12 months
  Assessment of target tumour local control defined as local suspicious growth under CT imaging at the originally ablated target tumour within or abutting the ablation zone.
Device user experience | Day of procedure
  Device user experience questionnaire completed at the time of the procedure by the investigator or physician performing the ablation.
Assessment of pulmonary function | 12 months
  Completion of Pulmonary Function Tests to assess pulmonary function.
Ablation ablative margin assessment | Discharge - Day 1
  Evaluation of the size of the ablation margin defined as the ablation beyond the borders of the tumor by CT imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Bartholomew's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No